CLINICAL TRIAL: NCT04546334
Title: The Effect of Erector Spinae Plane Block on the Relief of Pain of Post-herpetic Neuralgia: Randomized Controlled Study
Brief Title: Erector Spinae Plane Block in Post-herpetic Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 34043/08/20
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Postherpetic Neuralgia
Keywords: Herpes Zoster; Postherpetic neuralgia; Erector spina plane block
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The patients will be blinded to their groups and a sham block will be performed.
  * An anesthesia resident who will not participate in the study and have no subsequent rule in it will help in the preparation of local anesthetic mixtures under strict aseptic precautions.
  * An assistant nurse who will be blinded to the study groups and will have no subsequent rule in it will help in collection of the data of measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients will be subjected to the routine medical treatment of post herpetic neuralgia as controls (Pregabalin, acyclovir, and paracetamol) and sham erector spinae plane block
  Interventions: Drug: Medical treatment; Procedure: Sham Erector Spinae block
- Group B (Experimental): Patients will be subjected to erector spinae block by bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose) together with medical treatment.
  Interventions: Drug: Medical treatment; Procedure: Real Erector Spinae block
- Group C (Experimental): Patients that will be subjected to erector spinae block by bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose with the addition of MgSO4 (equivalent to 100 mg)) together with medical treatment.
  Interventions: Drug: Medical treatment; Procedure: Real Erector Spinae block with magnesium sulphate

INTERVENTIONS:
Drug: Medical treatment — routine medical treatment of post herpetic neuralgia as controls (Pregabalin, acyclovir, and paracetamol)
Procedure: Real Erector Spinae block — Ultrasound guided Erector spinae plane block with injection of local anesthetic bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose)
  Arms: Group B
Procedure: Real Erector Spinae block with magnesium sulphate — Ultrasound guided Erector spinae plane block with injection of local anesthetic bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose with the addition of MgSO4 (equivalent to 100 mg))
  Arms: Group C
Procedure: Sham Erector Spinae block — Ultrasound guided Erector spinae plane block with injection ofnormal saline
  Arms: Group A

SUMMARY:
This randomized clinical study will be carried out on 72 patients admitted to the pain clinic in Tanta University Hospitals with post-herpetic neuralgia.

Cases presenting to the Pain Clinic with acute pain due to postherpetic neuralgia in thoracic and/or lumbar dermatomes with numerical rating scale (NRS) of 6 or more and they will be randomly divided, using the closed envelop method, into three equal groups.

Group A (24 patients): Patients will be subjected to the routine medical treatment of post herpetic neuralgia as controls (Pregabalin, acyclovir, and paracetamol) and sham erector spinae plane block Group B (24 patients): Patients will be subjected to erector spinae block by bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose) together with medical treatment.

Group C (24 patients): Patients that will subjected to erector spinae block by bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose with the addition of MgSO4 (equivalent to 100 mg)) together with medical treatment.

Primary outcome will be the efficacy of pain relief Secondary outcome will be the frequency of pain and the consumption of analgesics.

DETAILED DESCRIPTION:
This comparative randomized controlled study will be conducted on 72 patients of both gender suffering from post-herpetic neuralgia and presented at Pain Clinics of Tanta University Hospitals for a period of 9 months (September 2020- June 2021) that will be started immediately after obtaining Ethical Committee approval. An informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

A total of 72 cases with post herpetic neuralgia will be included in the current study, and they will be randomly divided, using the closed envelop method, into three equal groups.

Group A (24 patients): Patients will be subjected to the routine medical treatment of post herpetic neuralgia as controls (Pregabalin, acyclovir, and paracetamol) and sham erector spinae plane block Group B (24 patients): Patients will be subjected to erector spinae block by bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose) together with medical treatment.

Group C (24 patients): Patients that will subjected to erector spinae block by bupivacaine (2 - 2.5 mg/kg, with a maximum of 175 mg/dose with the addition of MgSO4 (equivalent to 100 mg)) together with medical treatment.

* Management of the patients Before intervention, all cases will be subjected to complete history taking, physical examination, and routine laboratory and radiological investigations (if other causes rather than post herpetic neuralgia are suspected). Pre intervention pain will be evaluated by NRS and recorded for all cases.
* Measurements An assistant resident will help in obtaining and recording our measurements. All the patients will undergo regular follow up visits that will be arranged throughout the upcoming 3 months following injection as every week in the first month, then, every 2 weeks in the next two months.

  1. Demographic data: including age, gender, associated morbidities, and site of post-herpetic neuralgia.
  2. Duration of analgesia will be defined as the analgesia starting from the performance of the block until the first analgesic requirement or reporting a pain score of 4/10.(9)
  3. Frequency of pain
  4. Numerical rating score NRS (0- 10 metric score to assess the severity of pain where 0= no pain and 10 = severe pain)
  5. Dose of pregabalin consumed per day to relief pain
  6. Dose of other analgesics required to control pain.

ELIGIBILITY:
Inclusion Criteria:

* Cases presenting to the Pain Clinic with acute pain due to postherpetic neuralgia in thoracic and/or lumbar dermatomes with a numerical rating scale (NRS) of 6 or more.

Exclusion Criteria:

* Patients commenced on opioids for any other reason rather than postherpetic neuralgia
* Secondary bacterial infection at the site of injection
* Uncontrolled psychiatric illness
* Uncooperative patients
* Refusal to participate in the study
* Diagnosed or suspected coagulopathy
* Morbid Obese patients with BMI >50 kg/m2
* Known history of allergy to local anesthetics
* Platelet count less than 75,000/ cc

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-26 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
The efficacy of pain relief | within 3 months of theinjection
  Numerical rating score NRS (0- 10 metric score to assess the severity of pain where 0= no pain and 10 = severe pain)

SECONDARY OUTCOMES:
The frequency of pain | within 3 months of theinjection
  The number of pain attacks (pain score of 4 or more)

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, M.D, Principal Investigator — Tanta University
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: SAP, ICF
Time Frame: 6 months after approval of the publication of the trial.
Access Criteria: Contact the principal investigator